CLINICAL TRIAL: NCT05133258
Title: Measuring Antibiotic Solution Concentration at the Tympanic Membrane Following Self-administration by Patients With Chronic Suppurative Otitis Media
Brief Title: Antibiotic Concentration After Delivery to Middle Ear for Chronic Suppurative Otitis Media
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, James E. Saunders, Professor of Otology / Neurotology, Dartmouth-Hitchcock Medical Center
Other Study IDs: STUDY02001093
Record Dates: First submitted 2021-10-25; First posted 2021-11-24 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Chronic Suppurative Otitis Media
Keywords: csom; antibiotic resistance; chronic suppurative otitis media; ototopical ciprofloxacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Aspirates of middle ear fluid with be collected to investigate antibiotic delivery. Auricular aspirates will be analyzed by reverse-phase liquid chromatography with tandem mass spectrometry to determine concentrations of ciprofloxacin in the middle ear after standard-of-care antibiotic delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic Suppurative Otitis Media group: Enrolled subjects with persistent otorrhea due to CSOM and prescribed with standard of care (prescription for antibiotic drops from a pharmacy of their choice with specific written instructions for self-administration).
  Interventions: Other: Aspiration of middle ear fluid following standard-of-care delivery of ciprofloxacin and dexamethasone suspension

INTERVENTIONS:
Other: Aspiration of middle ear fluid following standard-of-care delivery of ciprofloxacin and dexamethasone suspension — Micro-aspirate of middle ear fluid will be taken from participants with a Juhn Tym-Tap specimen trap following standard-of-care delivery of ciprofloxacin 0.3% and dexamethasone 0.1% suspension. Samples will be analyzed to measure antibiotic concentration in the middle ear fluid.

SUMMARY:
The study team aims to elucidate the potential role of ototopical antibiotic concentration on outcomes in patients diagnosed with chronic suppurative otitis media (CSOM). Chronic suppurative otitis media (CSOM) is characterized by chronic inflammation of the middle ear with persistent discharge from a non-intact tympanic membrane. CSOM is notably associated with a significant burden of disease worldwide. Topical fluoroquinolones are first line therapy for CSOM and are advantageous as compared to oral or intravenous therapy in that these antibiotics avoid systemic side effects and have the potential to locally deliver high antibiotic concentrations, which were thought to be sufficient to overcome all bactericidal resistance to fluoroquinolones.

The investigators will measure antibiotic concentration in aspirates via liquid chromatography with tandem mass spectrometry (LC-MS/MS) from the middle ear of selected subjects with CSOM who are prescribed and instructed to self-administer ototopical ciprofloxacin. Enrolled subjects will be asked to return 3 to 10 days after initial visit to aspirate the middle ear and receive a follow-up evaluation. Furthermore, the subjects will be asked to keep logs of their medication use and to administer the ototopical medication one hour prior to their appointments. The measured ciprofloxacin concentrations will be correlated with clinical outcomes, primarily the time to symptom resolution. The guiding hypothesis is that patient self-administration of ciprofloxacin drops vary in antibiotic delivery with diluted concentrations significantly below the in vitro concentration of the prescribed solution and that these concentrations are below the bactericidal concentration of ciprofloxacin-resistant bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients greater than or equal to 18 years of age
* Diagnosis of Chronic Suppurative Otitis Media (CSOM)

Exclusion Criteria:

* Atypical presentation of CSOM or atypical anatomy of the ear
* Presence of additional ear pathophysiology beyond CSOM
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ten subjects will be accrued locally in the ENT clinic on 4F at tertiary care center Dartmouth-Hitchcock Medical Center in Lebanon, NH, using inclusion/exclusion criteria listed above.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Concentration of Ciprofloxacin | 3 to 10 days after initial visit
  Antibiotic Delivery to the Middle Ear will be measured by Ciprofloxacin concentration Relevant concentration range is 2000 ng/mL to 2,000,000 ng/mL, which are the minimum inhibitory concentration and theoretical maximum concentration, respectively. Measured through LC-MS/MS, aspirate collected 3-10 days after initial visit.

SECONDARY OUTCOMES:
Patient Compliance to Treatment as measured by Daily Compliance + Symptom Log | Starting after the initial visit, for 10 days
  The patient is given a medication and symptoms log to track administration of ototopical ciprofloxacin treatment (3 times per day for 10 days).
Persistence of Symptoms as measured by Daily Compliance + Symptom Log | Starting after the initial visit, for 10 days. Afterwards, weekly surveys to monitor symptoms for a maximum followup of 12 weeks.
  The patient is given a medication and symptoms log to track status of symptoms, which include ear discomfort, ear discharge, ear fullness, hearing changes, and "other."

CONTACTS AND LOCATIONS:
Overall Officials: James E Saunders, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT05133258/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT05133258/ICF_001.pdf